CLINICAL TRIAL: NCT04247659
Title: Study on the Relationship Between Asymmetric Vascular Sign of Cortex and Cerebral Edema and Prognosis of Massive Cerebral Infarction
Brief Title: Study on the Relationship Between Asymmetric Vascular Sign of Cortex and Prognosis in Massive Cerebral Infarction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, liuxiaoyun, Deputy director of neurology, The Second Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-P002
Record Dates: First submitted 2020-01-09; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Cerebral Infarction; Cerebral Edema
Keywords: massive cerebral infarction; asymmetric vascular sign of cortex; Sodium aescinate
MeSH Terms: conditions — Cerebral Infarction; Brain Edema | interventions — sodium aescinate; Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In the experimental group, sodium aescinate is added on the basis of conventional treatment(such as anti-platelet and improve circulation).The treatment course of sodium aescinate is 10 days,20mg/day.
  Interventions: Drug: sodium aescinate
- Control group (No Intervention): The control group will receive conventional treatment(anti-platelet and improve circulation) without sodium aescinate.

INTERVENTIONS:
Drug: sodium aescinate — The main mechanism of sodium aescinate includes anti - inflammatory, anti - exudate anti - oxygen free radical ,anti - edema increased venous tension.The treatment course of sodium aescinate is 10 days,20mg/day, intravenous infusion.
  Other Names: Sodium Aescinate for Injection
  Arms: Experimental group

SUMMARY:
Susceptibility weighted imaging (SWI) technology has developed in the decade which is being a kind of cerebrovascular disease diagnostic tools in the clinical application, especially for paramagnetic material (such as DNA hemoglobin and hemosiderin) has a high sensitivity.

The change of the signal on SWI bases on the change of local oxygenated hemoglobin content in the blood and deaeration hemoglobin content ratio, which can be used to indirectly reflect the hypoxia group oxygen intake fraction (OEF) and cerebral metabolic rate. When the intracranial vascular occlusion, corresponding responsibility vascular blood flow area of brain tissue will occur hypoperfusion, brain tissue will improve the compensation in accordance with its own OEF, causing ischemia area inside the venous drainage of deaeration hemoglobin content ratio increases and the hypointensity on SWI ,which display the asymmetric cortical vessel sign (ACVS). Studies have suggested that ACVS is more prone to early neurological deterioration and has a poor long-term outcome. After recanalization of ischemic stroke, the presence of equal CVS(return to normal) on SWI is associated with a good clinical outcome. In addition, the relationship between ACVS grade and collateral circulation in patients with acute ischemic stroke has been studied. For patients with massive cerebral infarction, the relationship between ACVS on SWI and the clinical prognosis of cerebral edema and cerebral hemodynamics is not completely clear. In this study, the clinical data of patients with massive cerebral infarction will be analyzed to explore the relationship between ACVS, cerebral edema , cerebral hemodynamic and clinical prognosis.

Sodium aescinate is widely used in cerebral edema caused by cerebral hemorrhage or cerebral infarction.The main mechanism of sodium aescinate is anti - inflammatory, anti - exudate, anti - oxygen free radical, anti - edema, increase vein tension, improve blood circulation and nerve protection. In this study, investigators will investigate whether the application of sodium aescinate had an effect on ACVS on SWI in patients with massive cerebral infarction. Plasma s100-β, procalcitonin, neutrophil count, serum fibronectin, and endothelin-1 could predict cerebral edema in patients with cerebral infarction, this study will analyze the relationship between these markers and ACVS on SWI in patients with massive cerebral infarction.

DETAILED DESCRIPTION:
Clinical data and plasma samples of patients diagnosed with massive cerebral infarction in the department of neurology of the second hospital of hebei medical university during 2020.1-2021.6 are collected.Clinical data include gender, age, TOAST classification, history of hypertension, diabetes and heart disease, head Computerized Tomography (CT), Magnetic Resonance Imaging(MRI), Diffusion-Weighted Imaging (DWI),Susceptibility weighted imaging SWI within 72 hours after onset, admission National Institute of Health stroke scale ( NIHSS) score, admission DWI-aspect score, Modified Rankin Scale (MRS) score on day 90 of onset.Venous blood will be taken within 72 hours of onset (and before the use of sodium aescinate) to detect serum s100-β, serum procalcitonin, plasma fibronectin, serum endothelin-1 by ELISA.The cortical vessel signs（CVSs）on SWI in the ischemic territory are classified as 'prominent' if there are more veins and/or larger veins with a greater signal loss than those in the opposite normal hemisphere, 'equal' if there are no significant differences in appearance of veins in the both cerebral hemispheres, and 'less' if the veins in the affected area are decreased compared to those in the normal cortex.

Patients with massive cerebral infarction to be included are randomly divided into experimental group and control group by random number table method.The experimental group is treated with sodium aescinate for injection on the basis of conventional treatment. The control group is not treated with sodium aescinate for injection.

This study will explore the relationship between asymmetric cortical vessel sign(ACVS) grade and baseline clinical data, serum factors associated with brain edema in patients with massive cerebral infarction.In addition,after 10 days of sodium aescinate injection, the CVS level of the experimental group will be compared with that of the control group.The difference of CVS grading before and after injection of sodium aescinate in the experimental group will be compared.Finally,the indexes with significance in single factor analysis will be screened out, and the factors related to prognosis of massive cerebral infarction will be further analyzed by multi-factor logistics regression.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Massive cerebral infarction within 72 hours from onset to admission
* Without other intracranial lesions or severe disease
* Agrees to participate in the study and sign the informed consent

Exclusion Criteria:

* Cerebral vascular malformation
* Cranial trauma and cranial surgery history
* With severe cardiac, hepatic and renal insufficiency
* With blood disorder, immune rheumatism (hormone abuse)
* Expected survival of less than 3 months
* Refuse to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-06-09 (Estimated); Study Completion 2021-09-09 (Estimated)

PRIMARY OUTCOMES:
The correlation between asymmetric cortical vessel sign(ACVS) and age | 2 hour
  To evaluate whether ACVS and age are related
The correlation between asymmetric cortical vessel sign(ACVS) and sex | 2 hour
  To evaluate whether ACVS and sex are related
The correlation between asymmetric cortical vessel sign(ACVS) and TOAST subtypes | 2 hour
  Classification of causes of stroke --TOAST classification include Large-artery atherosclerosis( LAA),Cardioembolism(CE) ,Small-artery occlusion(SAO),Stroke of other determined cause(ODC) and Stroke of undetermined cause(UND).
The correlation between asymmetric cortical vessel sign(ACVS) and smoking history | 2 hour
  To evaluate whether ACVS and smoking history are related
The correlation between asymmetric cortical vessel sign(ACVS) and NIHSS score at admission | 2 hour
  The NIHSS score is 0 to 42 points. The higher the score, the more severe the nerve damage.
The correlation between asymmetric cortical vessel sign(ACVS) and mRS on 90 day | 2 hour
  The mRs score is used to measure the recovery of neurological function in patients after stroke. The mRs score is 0 to 6 points. The higher the score, the worse the neurological function recovery.
The correlation between asymmetric cortical vessel sign(ACVS) and DWI ASPECT | 2 hour
  ASPECT is a scale suitable for evaluating ischemic changes in the supply area of the middle cerebral artery with a total score of 10.A score of 10 indicates no signs of ischemia, while a score of 0 indicates extensive ischemia in the middle cerebral artery
The correlation between asymmetric cortical vessel sign(ACVS) and midline shift | 2 hour
  To evaluate whether ACVS and midline shift are related
The correlation between asymmetric cortical vessel sign(ACVS) and offending stenosis | 2 hour
  To evaluate whether ACVS and offending stenosis are related
The correlation between asymmetric cortical vessel sign(ACVS) and serum factor S100-B | 2 hour
  In acute ischemic stroke, the astroglial protein S100B is released into peripheral blood, reaching maximum serum concentrations between day 2 and day 4, correlating with infarct size.
The correlation between asymmetric cortical vessel sign(ACVS) and serum factor procalcitonin | 2 hour
  Procalcitonin is a stronger predictor of long-term functional outcome and mortality in patients with ischemic stroke.
The correlation between asymmetric cortical vessel sign(ACVS) and cellular-fibronectin | 2 hour
  A high plasma cellular-fibronectin concentration at admission is associated with the development of m-MCA infarction with high sensitivity and specificity.
The correlation between asymmetric cortical vessel sign(ACVS) and serum factor endothelin - 1 | 2 hour
  endothelin - 1 may be a diagnostic marker for development of severe brain edema in patients with acute ischemic stroke.
Changes of aescinin on asymmetric cortical vessel sign (ACVS). | 2 hour
  This study investigates whether the application of sodium aescinate has an effect on ACVS on SWI in patients with massive cerebral infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyun Liu, Prf., Principal Investigator — The Second Hospital of Hebei Medical University
Locations (1):
- Second hospital of hebei medical university, Shijiazhuang, Hebei, China